CLINICAL TRIAL: NCT03342261
Title: Benefit of Direct-acting Antiviral Therapy in Hepatitis C Virus (HCV) Monoinfected and HIV-HCV Coinfected Patients With Mixed Cryoglobulinemia
Brief Title: Benefit of DAA Therapy in HCV Monoinfected and HIV-HCV Coinfected Patients With Mixed Cryoglobulinemia
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2017_002
Record Dates: First submitted 2017-11-07; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C, Chronic; Mixed Cryoglobulinemia
MeSH Terms: conditions — Hepatitis C, Chronic; Cryoglobulinemia, Familial Mixed | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCV patients with mixed cryoglobulinemia: HCV patients with or without HIV presenting a mixed cryoglobulinemia and treated with direct-acting antiviral agents
  Interventions: Drug: DAA treatment

INTERVENTIONS:
Drug: DAA treatment — Patients were treated with direct-acting antiviral (DAA) treatment for 12 or 24 weeks
  Other Names: Treatment with direct-acting antiviral agents

SUMMARY:
Mixed cryoglobulinemia (MC) is common in patients with chronic hepatitis C virus (HCV) infection. Direct-acting antiviral (DAA) regimens are today very effective with sustained virological response rates (SVR12) above 90%. The objective of this study was to investigate the impact of DAA therapy on cryoglobulin clearance in patients with HCV-associated MC.

DETAILED DESCRIPTION:
We focused on HCV patients with or without HIV with MC who had at least one cryoglobulin level assessment before and after DAA therapy and investigated the impact of DAA therapy on cryoglobulin clearance.

ELIGIBILITY:
Inclusion Criteria:

* hepatitis C virus (HCV) infected patients
* symptomatic or asymptomatic mixed cryoglobulinemia
* coinfected or not with HIV
* treated by direct-acting antiviral (DAA) treatment
* at least one cryoglobulin measurement before and after DAA

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV patients with mixed cryoglobulinemia
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Cryoglobulin level at the end of therapy | End of treatment (12 or 24 weeks)
  The primary outcome was the cryoglobulin level at the end of direct-acting antiviral treatment (week 12 or 24 according to treatment duration)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Zoulim, MD, PhD, Study Chair — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Croix-Rousse Hospital, Lyon, France

IPD SHARING:
Plan to Share IPD: No